CLINICAL TRIAL: NCT03817749
Title: The Effects of Exogenous Ketone Supplementation on Cardiovascular Function and Glucose Control
Brief Title: Ketone Supplementation, Glucose Control, and Cardiovascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: H18-02930
Record Dates: First submitted 2018-12-06; First posted 2019-01-25 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hyperglycemia, Postprandial; Overweight and Obesity; Diabetes Mellitus Risk
Keywords: Flow mediated dilation; Glucose control; Inflammation; Immune cell function; Cognition; Oxidative stress; Cardiovascular function
MeSH Terms: conditions — Hyperglycemia; Overweight; Obesity; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): * Participants will consume 20 g of an active oral exogenous ketone monoester supplement 15 minutes prior to each meal of the day for a 14-day period.
  * Pre-intervention (baseline) and post-intervention measurements will be obtained before and immediately after the 14-day period.
  * All meals will be provided throughout the supplementation period
  * Participants will wear a continuous glucose monitor for 6 consecutive days during the supplementation period.
  Interventions: Dietary Supplement: Exogenous ketone monoester
- Placebo (Placebo Comparator): Participants will consume a flavor matched placebo drink and undergo the same procedures described in the Experimental Arm
  Interventions: Dietary Supplement: Exogenous ketone monoester

INTERVENTIONS:
Dietary Supplement: Exogenous ketone monoester — Participants will consume 20g of the oral ketone monoester supplement 15 minutes prior to each meal of the day for 14 days. All meals will be provided throughout the 14-day supplementation period.
  Other Names: HVMN ketone monoester supplement

SUMMARY:
Post-prandial hyperglycemic excursions induce a cascade of deleterious effects on the body, including increased inflammation, production of reactive oxygen species, and impaired cardiovascular function. Ingestion of an exogenous oral ketone supplement blunts hyperglycemia in response to an oral glucose tolerance test. Accordingly, it is hypothesized that exogenous ketone supplement ingestion prior to a meal could be an effective strategy for blunting postprandial hyperglycemia. Therefore, the purpose of this study is to investigate the effect of short-term (14-days) pre-meal exogenous ketone supplementation on glucose control, cardiovascular function, inflammation, and oxidative stress in individuals at an elevated risk of type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Elevated waist circumference (>102 cm for males, >88 cm for females) and/or Obesity (BMI > 30 kg/m2) and/or Diagnoses of prediabetes based on A1C (5.7-6.4%) and/or fasting plasma glucose (5.6-6.9 mmol/l) using ADA criteria

Exclusion Criteria:

* Competitively trained endurance athlete
* Actively attempting to lose weight
* History of mental illness or existing neurological disease(s)
* Previous cardiovascular events (i.e., heart attack, stroke)
* Diagnoses of diabetes
* Hypoglycemia
* Irritable bowel syndrome or inflammatory bowel disease
* Taking medication that may interfere with insulin sensitivity
* Currently following a ketogenic diet or taking ketone supplements
* Unable to commit for 2 separate 14-day trials and unable to follow a controlled diet

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Glucose control | 2 hours after a meal
  Post-prandial glucose excursions will be measured by continuous glucose monitoring using the iPro2 CGM by Medtronic in both the active and placebo supplement conditions. Post-prandial glucose following breakfast, lunch, and dinner will be averaged together.

SECONDARY OUTCOMES:
Change from baseline flow mediated dilation at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Vascular function will be assessed by flow mediated dilation of the brachial artery using vascular ultrasound. A cuff will affixed on the forearm, distal to the brachial artery and will be inflated for 5 minutes. Flow mediation dilation will be measured over a 3-minute period following cuff release.
Change from baseline histone acetylation at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Histone H3 acetylation status will be quantified by flow cytometry using conjugated acetyl-histone H3 antibody specific for Lys9 (Pacific Blue 445) and the conjugated acetyl-histone H3 antibody specific for Lys14 (Alexa Fluor 488).
Change from baseline mitochondrial superoxide production at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Oxidative Stress will be measured by mitochondrial superoxide production in blood lymphocytes, monocytes, and neutrophils by flow cytometry using the MitoSOX red assay (ThermoFisher #M36008) and total intracellular ROS via the DCFDA assay (Sigma #D6883)
Change from baseline cognition (executive functions) at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Cognition will be assessed using a customized battery of psychometrically validated tests within the domain of executive functions using the iPad-based app BrainBaseline. The tests will be the Stroop test, task-switching test, digit-symbol substitution test, and the n-back test.
Change from baseline plasma glucose at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Venous blood samples will be taken and plasma glucose will be measured using a hexokinase method.
Change from baseline plasma insulin at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Venous blood samples will be taken and plasma insulin will be measured using a high-sensitivity human insulin ELISA.
Change from baseline plasma free fatty acids at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Venous blood samples will be taken and free fatty acids will be measured by colorimetric assay.
Change from baseline interleukin-1(IL)-1beta at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Mature IL-1beta secretion will be quantified by ELISA run in duplicate
Change from baseline caspase-1 activation at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Caspase-1 activation will be quantified by flow cytometry. The fluorescent inhibitor probe FAM-YVAD-FMK binds covalently to activated caspase-1 and emits at 530nm

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia, Okanagan., Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will share individual patient data (de-identified) with researchers upon request.

REFERENCES:
- [Derived] Walsh JJ, Caldwell HG, Neudorf H, Ainslie PN, Little JP. Short-term ketone monoester supplementation improves cerebral blood flow and cognition in obesity: A randomized cross-over trial. J Physiol. 2021 Nov;599(21):4763-4778. doi: 10.1113/JP281988. Epub 2021 Oct 4. PMID 34605026
- [Derived] Walsh JJ, Neudorf H, Little JP. 14-Day Ketone Supplementation Lowers Glucose and Improves Vascular Function in Obesity: A Randomized Crossover Trial. J Clin Endocrinol Metab. 2021 Mar 25;106(4):e1738-e1754. doi: 10.1210/clinem/dgaa925. PMID 33367782